CLINICAL TRIAL: NCT03171194
Title: A Phase I Safety Trial of Allogeneic Mesenchymal Stem Cells for Systemic Lupus Erythematosus
Brief Title: Pilot Trial of Mesenchymal Stem Cells for Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00061632
Record Dates: First submitted 2017-05-04; First posted 2017-05-31 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: System; Lupus Erythematosus
Keywords: Lupus; Stem Cell; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug: Low Dose Mesenchymal Stem Cells ( MSCs) (Experimental): Participants will receive a single IV infusion of Mesenchymal Stem Cells (MSCs) 1 x 10^6 cells/kg in Plasma-Lyte A solution. All participants will receive the infusion at the Baseline (Day 0) visit. All participants will continue on their standard-of-care therapy during the trial.
  Interventions: Drug: Low Dose Mesenchymal Stem Cells (MSCs)

INTERVENTIONS:
Drug: Low Dose Mesenchymal Stem Cells (MSCs) — Mesenchymal stromal/stem cells (MSCs) are cells that can be derived from umbilical cords, bone marrow, adipose tissue, and dental pulp, among other sites. MSCs have the ability to mediate a range of immuno-modulatory actions for both the innate and adaptive immune systems.

SUMMARY:
The purpose of this study is to evaluate the safety of mesenchymal stromal cells (MSCs) obtained from umbilical cords for the treatment of adults with active systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
This open label trial will evaluate the safety of allogeneic MSCs for the treatment of adults with moderate to severely active systemic lupus erythematosus (SLE). MSCs will be derived from healthy donor umbilical cord cells and 1 dose of MSCs will be tested. MUSC has a good manufacturing practice (GMP) quality Clean Cell Facility to ensure the quality and safety of the MSCs prior to infusing into study participants. The goal of this study is to determine the safety of MSC infusion in patients with SLE when added to standard of care for SLE.

The MSCs used in this trial are cells that are obtained from the umbilical cords of healthy donors having an elective Caesarean section and who have been screened to be sure that they are free of any infectious diseases. These investigational cells will be collected and processed so that they can be used as an infusion treatment. An infusion is when a drug (in this case the MSCs) is administered directly into the blood stream via a vein, usually located in the arm or hand. All participants will receive standard of care and their safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years old, male or female, of any race
* Definite SLE by meeting either SLICC or ACR Classification Criteria for SLE
* Evidence of a positive ANA (≥1:80 titer) or positive dsDNA antibody test within 6 months of screening
* Clinically mild to moderately active SLE determined by SLEDAI score ≥4 and ≤10 at screening, despite SOC therapy
* If the patient has BILAG A or two BILAG Bs in the renal organ system, he/she must have completed at least 6 months of therapy with either mycophenolate mofetil or cyclophosphamide for the current episode of nephritis
* Able and willing to give written informed consent

Exclusion Criteria:

* Active CNS lupus affecting mental status
* Active lupus nephritis requiring dialysis
* Laboratory exclusions: eGFR <30, WBC <2.0/mm3, hemoglobin <8 g/dL, platelet count <30,000/mm3, liver enzymes AST or ALT >4 times upper limit normal; Positive testing for HIV, hepatitis B or hepatitis C
* History of malignant neoplasm within the last 3 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix
* Pregnant or breast feeding; males or females not willing to use adequate contraception
* History of renal transplantation
* Herpes zoster within the past 90 days or any infection requiring hospitalization or intravenous antibiotics within the past 60 days
* Clinically significant EKG or chest X-ray abnormalities
* Any other medical condition, related or unrelated to SLE, that in the opinion of the investigator would render the patient inappropriate or too unstable to complete study protocol
* Use of prednisone >0.5 mg/kg/day (or equivalent corticosteroid) within 1 month of Baseline visit
* Change or addition to immunosuppressant regimen within 3 months of Baseline visit (except corticosteroids); Use of other experimental therapeutic agents within 3 months of Baseline visit
* Having received belimumab within 3 months of Baseline, or having received rituximab or other B cell depleting biologic therapy within 6 months of Baseline.
* Comorbidities requiring corticosteroid therapy
* Current substance abuse or recent (within 60 days) history of substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Frequency of Grade 3 or higher adverse events | Week 24
  The primary outcome measure is the frequency of Grade 3 or higher adverse events (AEs) experienced by participants at or prior to Week 24.

SECONDARY OUTCOMES:
Frequency of All Adverse Events | Baseline to Week 52
  Frequency of all adverse events (AEs) including any serious AEs (SAEs) at or prior to Week 52.
Change in Disease Activity | Baseline to Week 24
  Change in SLE disease activity between Baseline and Week 24 measured by change in SLEDAI score and change in prednisone dose.
Change in Patient Reported Outcomes - Life | Baseline to Week 24
  Changes between Baseline and Week 24 in patient-reported quality of life
Change in Patient Reported Outcomes - Fatigue | Baseline to Week 24
  Changes between Baseline and Week 24 in patient-reported measures of fatigue.
Change in Patient Reported Outcomes - Pain | Baseline to Week 24
  Changes between Baseline and Week 24 in patient-reported measures of pain.
Change in Patient Reported Outcomes - Depression | Baseline to Week 24
  Changes between Baseline and Week 24 in patient-reported measures of depression.
Change in Disease Biomarkers - Cellular | Baseline to Week 24
  Changes between Baseline and Week 24 in cellular markers of inflammation and autoimmunity. Mechanistically, the study will test the hypothesis that MSC infusions in patients with active SLE will increase Treg numbers via enhancing TGF-beta activity while decreasing T and B cell effector subsets.
Change in Disease Biomarkers - Serum | Baseline to Week 24
  Changes between Baseline and Week 24 in serum markers of inflammation and autoimmunity. Mechanistically, the study will test the hypothesis that MSC infusions in patients with active SLE will increase Treg numbers via enhancing TGF-beta activity while decreasing T and B cell effector subsets.

CONTACTS AND LOCATIONS:
Overall Officials: Diane L. Kamen, MD, MSCR, Study Chair — Medical University of South Carolina
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamen DL, Wallace C, Li Z, Wyatt M, Paulos C, Wei C, Wang H, Wolf BJ, Nietert PJ, Gilkeson G. Safety, immunological effects and clinical response in a phase I trial of umbilical cord mesenchymal stromal cells in patients with treatment refractory SLE. Lupus Sci Med. 2022 Jul;9(1):e000704. doi: 10.1136/lupus-2022-000704. PMID 35820718